CLINICAL TRIAL: NCT03494140
Title: Viscontour® Serum Med in Hydration of Facial Skin
Status: Completed | Type: Observational
Sponsor: TRB Chemedica AG (Industry)
Responsible Party: Sponsor
Other Study IDs: VISCH-PMCF-DE-2016-09
Record Dates: First submitted 2018-03-26; First posted 2018-04-11 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Sodium Hyaluronate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Viscontour® Serum Med — Viscontour® Serum Med is a CE-certified preservative-free isotonic solution containing 5.0 mg sodium hyaluronate.

SUMMARY:
The objective of this study is to confirm the clinical safety and efficacy of Viscontour® Serum Med in the hydration of facial tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Females ≥ 18 years of age and in good general health condition
2. Signed informed consent
3. Existing Viscontour® Serum Med recommendation (i.a. for hydration, soothing, nourishing and refreshing the complexion and for use in combination with a day cream)

Exclusion Criteria:

1. Known hypersensitivity to one of the Viscontour® Serum Med components
2. Known pregnancy or lactating females
3. Subjects not capable of contracting and of understanding the nature, risks, significance and implications of the clinical investigation and unable to form a rational intention in the light of these facts
4. Subjects unable to understand informed consent or having a high probability of non compliance to the study procedures and / or non completion of the study according to investigator's judgement (e.g. illiteracy, insufficient knowledge of local language)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a Viscontour® Serum Med therapy recommendation (i.a. for hydration, soothing, nourishing and refreshing the complexion and for use in combination with a day cream)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2018-08-18 (Actual); Study Completion 2018-08-18 (Actual)

PRIMARY OUTCOMES:
Change of Skin Parameters compared to Baseline | 20 Minutes, Day 7 and Day 28
  Routine Evaluation of the Overall Skin Condition
Change of Subjective Therapy Evaluation (Questionnaire) compared to Baseline | 20 Minutes, Day 7 and Day 28
Incidence of Treatment-Emergent Adverse Events | Up to Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Praxis Dr. Dirk Gröne, Berlin, Germany